CLINICAL TRIAL: NCT05994690
Title: An Open Label Complex Clinical Trial in Newly Diagnosed Pediatric de Novo AML Patients - a Study by the NOPHO-DB-SHIP Consortium, Master Protocol
Brief Title: CHIP-AML22/Master: An Open Label Complex Clinical Trial in Newly Diagnosed Pediatric de Novo AML Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-504999-25-00
Record Dates: First submitted 2023-07-25; First posted 2023-08-16 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard arm Rc (Active Comparator): 3 consolidation courses (HAM + HA3E + FLA)
  Interventions: Drug: Standard Intervention Rc
- Investigational arm Rc (Experimental): 2 consolidation courses (HAM + FLA)
  Interventions: Drug: Investigational Intervention Rc
- Standard arm Ri (Active Comparator): No addition om gemtuzumab ozogamicin (GO) to the first induction course of CD33-positive AML
  Interventions: Drug: Standard Intervention Ri
- Investigational arm Ri (Experimental): Addition om gemtuzumab ozogamicin (GO) to the first induction course of CD33-positive AML
  Interventions: Drug: Investigational Intervention Ri

INTERVENTIONS:
Drug: Standard Intervention Rc — 3 consolidation courses (HAM + HA3E + FLA)
  Arms: Standard arm Rc
Drug: Investigational Intervention Rc — 2 consolidation courses (HAM + FLA)
  Arms: Investigational arm Rc
Drug: Standard Intervention Ri — No addition of GO to first induction course
  Arms: Standard arm Ri
Drug: Investigational Intervention Ri — Addition of GO to first induction course
  Arms: Investigational arm Ri

SUMMARY:
The CHIP-AML22 Master protocol has the overall aim of increasing the cure rate in newly diagnosed pediatric de novo AML patients, while avoiding unnecessary toxicity.

DETAILED DESCRIPTION:
This is a master protocol comprising a complex clinical trial with a stratification approach to allocate patients to randomized studies described in the master protocol or linked trials.

The overarching objective of the CHIP-AML22 study is to improve event-free survival (EFS) in children and adolescents with AML, as compared to NOPHO-DBH 2012.

The consortium strives to achieve the overarching aim by:

1. Avoiding unnecessary toxicity. This will be investigated in a randomized setting (non-inferiority) by omitting a third standard-of-care consolidation course for standard-risk patients (4 versus 5 courses of chemotherapy).
2. Introducing quizartinib as FLT3-inhibitor in addition to the first three sequential chemotherapy courses for all patients with FLT3-ITD/NPM1wt, and as post-SCT continuation treatment for the subset of patients that have MRD ≥0.1% after course 1 or at any time-point later on (historical comparison, higher efficacy).
3. Refining risk-group adapted treatment, by classifying patients with KMT2A-rearrangement (except KMT2A/MLLT3) and MRD≥0.1% in BM after course 1 as high-risk (historical comparison, higher efficacy), as well as patients with the RAM-phenotype and/or CBFA2T3::GLIS2 fusion (historical comparison, higher efficacy). High-risk (non-FLT3-ITD/NPM1wt patients) will also be concluded for patients having ≥15% leukemic cells in BM after course 1, or ≥0.1-5% after course 2. Refractory disease will be defined as ≥5% leukemic cells in bone marrow after 2 courses of induction treatment, or disease elsewhere, or both.
4. Recommending the use of the cardioprotective drug dexrazoxane in all courses incorporating an anthracycline or mitoxantrone (exploratory objective, no statistical design), with the aim to prevent cardiotoxicity.
5. To assess if adding gemtuzumab ozogamicin to the first induction course results in better anti-leukemic efficacy in CD33-positive AML patients. Children with FLT3-ITD/NPM1wt are not eligible for this randomization.
6. To explore health-related Quality of Life during and after completion of treatment by using short questionnaires (exploratory objective, no statistical design).

ELIGIBILITY:
General inclusion criteria for CHIP-AML22/Master:

Patients are eligible for the study if they fulfil all four criteria below:

1. Newly diagnosed AML as defined by the diagnostic criteria in section 8.1. Note that different blast thresholds may apply for different genetic abnormalities in case of low blast percentages. The origin of AML must be de novo (not secondary to bone marrow failure or therapy-related).
2. Age ≥ day and ≤18 years old at initial diagnosis.
3. Written informed consent/assent from patients and/or from parents or legal guardians for minor patients, according to local law and regulations. Informed consent should ideally be obtained before day 7 of induction course 1, as patients that are eligible for the linked quizartinib trial should be enrolled before the end of induction course 1, and in view of the planned Mylotarg® randomisation. Thus, standard of care diagnostics and induction treatment may be started before informed consent has been obtained.
4. Able to comply with scheduled follow-up and with management of toxicity.

Additional inclusion criteria for Ri randomization

1. CD33 positivity of leukemic blasts as measured by flow cytometry at diagnosis (bone marrow aspirate and/or peripheral blood).
2. Informed consent for participation in randomization Ri

Additional inclusion criteria for Rc randomization

1. Patients included in the CHIP-AML22 protocol and stratified to Standard Risk Group according to the stratification algorithm of the protocol
2. Informed consent for participation in randomization Rc

General exclusion criteria for CHIP-AML22/Master

Patients are excluded if any of the criteria below are present:

1. Previous chemotherapy or radiotherapy. This includes patients with therapy-related AML after previous cancer therapy. These patients may be treated according to the master protocol but will not be part of the formal study population, and data of these patients will not be collected.
2. Patients with a (known) germline predisposition for bone marrow failure, like Fanconi anemia.
3. Myeloid Leukemia of Down syndrome (ML-DS). Patients with ML-DS are recommended to be treated according to the international ML-DS protocol. Patients with AML and DS older than 5 years who often lack GATA1 mutation and do not have typical myeloid leukemia of DS may be treated according to the master protocol but will not be part of the formal study population, hence data of these patients will not be collected.
4. Acute promyelocytic leukemia (APL).
5. Myelodysplastic syndrome (MDS).
6. Juvenile Myelomonocytic Leukemia (JMML).
7. Known intolerance to any of the chemotherapeutic drugs in the protocol.
8. Evidence of cardiac dysfunction (shortening fraction below 28%).
9. Pregnant or lactating patients, or sexually active female patients of childbearing potential not willing to use an highly effective method of contraception for the duration of study therapy and up to 7 months after the completion of all study therapy.
10. Sexually active, fertile male patients, not willing to use an effective method of contraception, for the duration of study therapy, and up to 6 months after the completion of all study therapy.
11. Concomitant administration of any other experimental drug under investigation, or concurrent treatment with any other anti-cancer therapy other than specified in this protocol or in one of the trials linked to this Master protocol, is not allowed.
12. Patients who in the opinion of the investigator, may not be able to comply with the study requirements of the study.
13. Patients with known active hepatitis B, hepatitis C, or HIV infection.
14. Patients for whom informed consent was not obtained.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 905 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Overarching primary objective | 5 years
  Event Free Survival (EFS)
Primary objective Randomisation Consolidation | 5 years
  Disease Free Survival (DFS)
Primary objective Randomisation Induction | 5 years
  MRD <0.1% leukemic cells in the BM

SECONDARY OUTCOMES:
Overarching secondary objective - efficacy 1 | 8 months
  • Bone marrow blast counts by morphology and multicolor flow cytometry (MFCM) after course #1 and #2 and before allo-SCT
Overarching secondary objective - efficacy 2 | 3 months
  ORR (CR, CRp, and CRi) and morphologic leukemia-free state (MLFS) rates after course #1 and #2;
Overarching secondary objective - efficacy 3 | 8 months
  MRD negativity after course #1 and #2 and before allo-SCT
Overarching secondary objective - efficacy 4 | 8 months
  Absolute MRD levels after course #1 and #2 and before allo-SCT
Overarching secondary objective - efficacy 5 | 5 years
  • OS
Overarching secondary objective - efficacy 6 | 5 years
  • DFS
Overarching secondary objective - efficacy 7 | 5 years
  • CIR
Overarching secondary objective - toxicity 1 | 5 years
  • Cumulative toxicity, defined as the total of all grades AEs over time, which are graded by NCI CTCAE version 5.0.
Overarching secondary objective - toxicity 2 | 5 years
  • NRM.
Secondary objective Randomisation consolidation - safety 1 | 8 months
  • Cumulative toxicity, defined as the total of grade ≥3 AESIs over time, which are graded by NCI CTCAE version 5.0.
Secondary objective Randomisation consolidation - safety 2 | 5 years
  • NRM.
Secondary objective Randomisation consolidation - healthcare resources | 1 year
  Cumulative Hospitalized Days
Secondary objective Randomisation consolidation - efficacy 1 | 5 years
  • OS
Secondary objective Randomisation consolidation - efficacy 2 | 5 years
  • CIR

CONTACTS AND LOCATIONS:
Overall Officials: Gertjan Kaspers, Prof. Dr., Study Chair — Pediatric Oncologist; Michel Zwaan, Prof. Dr., Study Director — Head Trial and Data Center
Locations (1):
- Princess Máxima Center for pediatric oncology, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be used to generate a publication
Supporting Information: CSR
Time Frame: Primary CSRs may be completed earlier when the primary objective is completed and may be followed by a final CSR not later than 6 months after the end of the trial.
Access Criteria: A summary of the study results will be made public via clinicaltrials.gov as well as to Ethical committees/ Health Authorities and all participating patients by providing them through their treating physicians a patient letter with a summary of the results.